CLINICAL TRIAL: NCT03533374
Title: Clinical Validation of Criteria for Identification of Epileptiform Electroencephalography Discharges in Sensor Space and Source Space
Brief Title: Validation of Criteria for Identification of Epileptiform Discharges in EEG Recordings of Patients With Epilepsy
Acronym: CIED
Status: Completed | Type: Observational
Sponsor: Sándor Beniczky (Other)
Collaborators: Aarhus University Hospital (Other); Central Denmark Region (Other); Filadelfia Epilepsy Hospital (Other); University Health Network, Toronto (Other); University Hospital Erlangen (Other); Oslo University Hospital (Other)
Responsible Party: Sponsor-Investigator, Sándor Beniczky, professor, Aarhus University Hospital
Organization: Aarhus University Hospital (Other)
Other Study IDs: CIED
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2019-07

CONDITIONS: Epilepsy; Non-Epileptic Seizure
Keywords: Accuracy; Inter-ictal EEG Discharges; Inter-rater agreement; Long Term Monitoring; Sensitivity; Sharp transients; Specificity; Source Space; Voltage maps
MeSH Terms: conditions — Epilepsy; Seizures; Hypersensitivity | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with epileptic seizures: Electroencephalogram (EEG) and visual evaluation
  - Electroencephalogram (EEG) was recorded using Nicolet-One system, and the standard 25-electrode array. Recordings with sharp transients are inspected by experts (physicians).
  Interventions: Diagnostic Test: Electroencephalogram (EEG) and visual evaluation
- Patients with non-epileptic seizures: Electroencephalogram (EEG) and visual evaluation
  - Electroencephalogram (EEG) was recorded using Nicolet-One system, and the standard 25-electrode array. Recordings with sharp transients are inspected by experts (physicians).
  Interventions: Diagnostic Test: Electroencephalogram (EEG) and visual evaluation

INTERVENTIONS:
Diagnostic Test: Electroencephalogram (EEG) and visual evaluation — Electroencephalogram (EEG) was recorded using Nicolet-One system, and the standard 25-electrode array. Recordings with sharp transients are inspected by experts (physicians).

SUMMARY:
Electroencephalography (EEG) records electric activity of the brain using electrodes placed on the scalp. EEG is an important tool in the diagnostic work-up of patients with epilepsy. Specific types of sharp EEG discharges (epileptiform discharges) are associated with patients with epilepsy.

The International Federation of Clinical Neurophysiology (IFCN) has recently published a set of six operational criteria for identifying epileptiform discharges. At least four criteria need to be present in order to classify a discharge as epileptiform. These criteria are largely based on expert opinion and have not been validated yet. It is not clear what the sensitivity and specificity of these criteria are, and which combination of these criteria are optimal. Each criterion is based on visual assessment. However, it is not known what the inter-rater agreement of these criteria are.

EEG is traditionally inspected in sensor space, i.e. in the recording channels. Advances in signal analysis made possible reconstructing the electric currents in the regions of the brain generating them, and displaying the signals in the source space, instead of the sensor space.

The objectives of this study are: to determine the inter-rater agreement of the IFCN criteria by visual analysis in sensor space, to determine the combination of criteria with the best accuracy (sensitivity and specificity) and assess the accuracy of evaluating the discharges in source space.

The raters will analyze EEG recordings from 100 patients, from two groups: consecutive patients with epilepsy and consecutive patients with non-epileptic paroxysmal episodes. EEG was recorded during long-term video-EEG monitoring. As reference standard, the investigators used the evaluation of the patients´ habitual clinical episode. The performance of the criteria in sensor-space and the analysis in source space will be compared with the unrestricted expert scorings.

DETAILED DESCRIPTION:
Epilepsy affects 50 million people of all ages. It is the most common neurologic disorder across the lifespan, and has been found to be associated with an increased risk of mortality compared to the general population.

EEG is an important tool in the diagnostic work-up of patients with suspected epilepsy. The presence of epileptiform EEG discharges (EDs) confirm the diagnosis and provides important information that helps in classifying epilepsy.

EDs are visually identified by experts with training in reading EEG. Although EDs were defined in the previous edition of the IFCN glossary of terms, that definition was conceptual, and the inter-rater agreement for identifying EDs was only moderate. Recently, the IFCN suggested the following operational definition for EDs: Transients distinguishable from background activity with a characteristic morphology; EDs have to fulfill at least 4 of the following 6 criteria:

1. Di- or tri-phasic waves with sharp or spiky morphology (i.e. pointed peak).
2. Different wave-duration than the ongoing background activity: either shorter or longer.
3. Asymmetry of the waveform: a sharply rising ascending phase and a more slowly decaying descending phase, or vice versa.
4. The transient is followed by an associated slow after-wave.
5. The background activity surrounding epileptiform discharges is disrupted by the presence of the epileptiform discharges.
6. Distribution of the negative and positive potentials on the scalp suggests a source of the signal in the brain, corresponding to a radial, oblique or tangential orientation of the source. This is best assessed by inspecting voltage maps constructed using common-average reference.

However, these criteria are largely based on expert opinion. Data from clinical validation studies are lacking, thus it is not known what the sensitivity and specificity of these methods are. The threshold of four fulfilled criteria was arbitrary, and it is not sure whether it yields the optimal accuracy (sensitivity and specificity). Furthermore, since each criterion is based on visual evaluation, it is not known whether all experts would reach the same conclusion.

The IFCN criteria were developed for identifying EDs using the traditional way of inspecting EEG, in the channels of the recording electrodes (sensor space). However, advances in signal analysis made possible to reproduce the electric currents in the brain regions, using a spatial filtering method (source space).

The objective of this study are:

1. To determine the inter-rater agreement for the IFCN criteria
2. To determine the number of criteria and their combination that yields the highest diagnostic accuracy
3. To determine the accuracy of identifying EDs in source space. Raters with experience in clinical EEG will inspect 100 anonymized EEG samples, from consecutive patients with epilepsy and consecutive patients with non-epileptic paroxysmal episodes. All 100 patients have a reference standard for their condition, derived from analysis of their video-EEG recordings of their habitual clinical episode. Patients with both focal and generalized epilepsy, as well as non-epileptic paroxysmal episodes (psychogenic non-epileptic seizures, sleep-disorders, movement disorders, convulsive syncope) are included.

Each EEG sample contains a sharp transient that is either epileptiform or not. EEGs were recoded using the IFCN electrode array of 25 electrodes (including the ones in the inferior temporal chain).

The samples were randomized twice, resulting in two series containing the same set of 100 samples, though with different codes and in different order of presentation. The raters will inspect the two series separately. In the first session the raters will inspect samples in sensor space, using traditional EEG montages (longitudinal and transversal bipolar; common average) and voltage maps. For each sample, they will score the presence or absence of each IFCN criterion. In the second session, the raters will inspect the EEG samples in source space and voltage maps, and will conclude on the presence / absence of EDs.

The performance of these methods will be compared with unrestricted scorings based on the experts´ evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who underwent long-term video-EEG monitoring
2. Patients who had at least one habitual episode (seizure) recorded on video and EEG.
3. Patients with sharp transients.
4. For patients with epilepsy: the interictal (epileptiform) sharp transients are concordant with the ictal recording

Exclusion Criteria:

Patients with both epileptic seizures and non-epileptic seizures (paroxysmal episodes).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patient with epilepsy and patient with non-epileptic seizures (paroxysmal episodes)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Epileptic Seizures; Patients With Non-epileptic Seizures: Electroencephalogram (EEG) and visual evaluation
  - Electroencephalogram (EEG) was recorded using Nicolet-One system, and the standard 25-electrode array. Recordings with sharp transients are inspected by experts (physicians).
  Electroencephalogram (EEG) and visual evaluation: Electroencephalogram (EEG) was recorded using Nicolet-One system, and the standard 25-electrode array. Recordings with sharp transients are inspected by experts (physicians).
Period: Overall Study
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures
Started | 54 | 46
Completed | 54 | 46
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures | Total
Number analyzed (Participants) | 54 | 46 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.5 (18.9) | 37.6 (19.7) | 34.8 (19.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 35 | 60
  Male | 29 | 11 | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 54 | 46 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Inter-rater Agreement of the International Federation of Clinical Neurophysiology (IFCN) Criteria (Cut-off=4) in Sensor Space and of Detection of Epileptiform Discharges (EDs) in Source Space
Description: Inter-rater agreement of IFCN criteria (cut-off=4) in sensor space and of detection of EDs in source space was calculated using Gwet´s Agreemen Coefficient (AC1).
  We calculated Gwet's coefficients of agreement AC1 for beyond chance agreement, because, compared with Cohen's Kappa, the Gwet's agreement coefficient is less affected by prevalence and marginal probability and thereby avoids the problem known as the "paradoxes of kappa". Strength of agreement beyond chance was interpreted according to Landis and Koch criteria: poor (<0), slight (0·01-0·20), fair (0·21-0·40), moderate (0·41-0·60), substantial (0·61-0·80), and almost perfect (0·81-1·00).
Time Frame: 1 year
Measure: Number (95% Confidence Interval); unit: AC1 - agreement coefficient
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures
Number analyzed (Participants) | 54 | 46
AC1 - agreement coefficient | 0.61 [0.53 to 0.69] | 0.59 [0.51 to 0.68]

2. Primary Outcome: Sensitivity and Specificity IFCN Criteria (Cut-off=4)
Description: This is a diagnostic study, hence sensitivity and specificity must be calculated from different groups: sensitivity form the group of patients with epilepsy and specificity from the gruoup of patients who do not have epilepsy.
  Sensitivity: the percentage of patients with abnormal index test (true positives) among patients with epilepsy.
  Specificity: the percentage of patients with normal index test (true negatives) among patients who do not have epilepsy.
Time Frame: 1 year
Population: Sensitivity is calculated in the epileptic group and specificity in the non-epileptic group.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures
Number analyzed (Participants) | 54 | 46
percentage | 96.3 [87.3 to 99.6] | 84.8 [71.1 to 93.7]

3. Primary Outcome: The Sensitivity and Specificity of Detecting EDs in Source-space
Description: This is a diagnostic study, hence sensitivity and specificity must be calculated from different groups: sensitivity form the group of patients with epilepsy and specificity from the group of patients who do not have epilepsy.
  Sensitivity: the percentage of patients with abnormal index test (true positives) among patients with epilepsy.
  Specificity: the percentage of patients with normal index test (true negatives) among patients who do not have epilepsy.
Time Frame: 1 year
Population: Sensitivity is calculated in the epileptic group and specificity in the non-epileptic group.
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures
Number analyzed (Participants) | 54 | 46
percentage | 85.2 [72.9 to 93.4] | 95.7 [85.2 to 99.5]

ADVERSE EVENTS:
Time Frame: Adverse Events were not monitored/assessed. Not applicable - this is a non-invasive diagnostic test.
Description: Adverse Events were not monitored/assessed. The procedure involved analysis of already recorded signals. Mortality risk and adverse events are not applicable in this diagnostic context.
Arm/Group | Patients With Epileptic Seizures | Patients With Non-epileptic Seizures
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-12-31): https://cdn.clinicaltrials.gov/large-docs/74/NCT03533374/Prot_000.pdf